CLINICAL TRIAL: NCT04255056
Title: The Effect of Pyrotinib in Breast Cancer Patients With Poor Response to the Neoadjuvant Treatment of Trastuzumab Combined With Pertuzumab: A Single-center Phase II Clinical Study
Brief Title: Pyrotinib in Breast Cancer Patients With Poor Response to the Neoadjuvant Treatment of Trastuzumab and Pertuzumab
Acronym: PRETTY
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xu fei, Associate Chief Physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSU-CSCO-2020
Record Dates: First submitted 2020-02-02; First posted 2020-02-05 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib (Experimental): Eligible patients will receive four cycles of epirubicin and cyclophosphamide combined with pyrotinib.
  Pyrotinib is administered orally at 400 mg daily from day 1 of the first cycle to day 21 of the fourth cycle or to the day of surgery, within 30 minutes after breakfast.
  Epirubicin (90 mg/m2), intravenously, every 21 days. Cyclophosphamide (600 mg/m2), intravenously, every 21 days.
  Interventions: Drug: Pyrotinib

INTERVENTIONS:
Drug: Pyrotinib — Pyrotinib is administered orally at 400 mg daily from day 1 of the first cycle to day 21 of the fourth cycle or to the day of surgery, within 30 minutes after breakfast.
  Epirubicin (90 mg/m2), intravenously, every 21 days. Cyclophosphamide (600 mg/m2), intravenously, every 21 days.
  Other Names: epirubicin; cyclophosphamide

SUMMARY:
Pathological complete remission (pCR) after neoadjuvant therapy in HER2-positive early breast cancer patients is closely related to disease-free survival (DFS) and overall survival (OS), which makes pCR an important evaluation indicator of recurrence risk. Trastuzumab combined with pertuzumab is a new standard targeted treatment regimen for HER2-positive early breast cancer. However, there are still quite a few patients who do not reach PCR. For these patients, current guidelines recommend the use of TDM-1 for intensive treatment after surgery, although a significant number of patients still have recurrence or metastasis. Besides, TDM-1 is unavailable in China. Pyrotinib has been approved for HER2-positive breast cancer patients who have previously failed after the treatment of trastuzumab. The investigators intend to conduct this phase II clinical study. Patients with poor response to the standard neoadjuvant treatment regimen of trastuzumab combined with pertuzumab are enrolled. These patients receive pyrotinib to observe that whether pCR has been improved. The investigators aim to explore the effect of pyrotinib in patients with poor response to standard dual-target neoadjuvant therapy, and further explore the improvement of neoadjuvant treatment strategy in HER2 positive early stage breast cancer patients.

DETAILED DESCRIPTION:
Breast cancer is the most common malignant tumor in Chinese women, with 20% to 30% HER2 overexpression. Pathological complete remission (pCR) after neoadjuvant therapy in HER2-positive early stage breast cancer patients is closely related to disease-free survival (DFS) and overall survival (OS), which makes pCR an important evaluation indicator of recurrence risk. Trastuzumab combined with pertuzumab is a new standard targeted treatment regimen for HER2-positive early breast cancer, with overall pCR rate of 57% to 66%. However, there are still quite a few patients who do not reach PCR after treatment in clinical practice. For patients who do not reach pCR with neoadjuvant therapy, current guidelines recommend the use of TDM-1 for intensive treatment after surgery, but even with TDM-1, a significant number of patients still have recurrence or metastasis. Besides, TDM-1 is currently unavailable in China. Pyrotinib has been approved for HER2-positive breast cancer patients who have previously failed after the treatment of trastuzumab. The investigators intend to conduct this single-arm, single-center phase II clinical study. Patients with poor response to the standard neoadjuvant treatment regimen of trastuzumab combined with pertuzumab are enrolled. These patients receive pyrotinib to observe that whether pCR has been improved after the replacement of targeted treatment regimen. The investigators aim to explore the effect of pyrotinib in patients with poor response to standard dual-target neoadjuvant therapy, and further explore the improvement of neoadjuvant treatment strategy in HER2 positive early stage breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged ≥ 18 years and ≤ 75 years;
2. ECOG score 0-1;
3. HER2-overexpressing breast cancer confirmed by immunohistochemical (IHC) analysis or in situ hybridization (ISH).
4. The patient has received at least 3 cycles of neoadjuvant therapy with trastuzumab combined with pertuzumab and the clinical response is SD or PD (according to RECIST version 1.1) evaluated with breast MRI/CT/ultrasound.
5. Known hormone receptor status (ER and PgR);
6. The function of the main organs must meet the following requirements： 1) Blood routine: Neutrophil (ANC) ≥1.5 × 10^9 / L; Platelet count (PLT) ≥90 × 10^9 / L; Hemoglobin (Hb) ≥90 g / L; 2) Blood biochemistry: Total bilirubin (TBIL) ≤ upper limit of normal value (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 × ULN; Alkaline phosphatase ≤ 2.5 × ULN; Urea nitrogen (BUN) and creatinine (Cr) ≤ 1.5 × ULN; 3) Cardiac ultrasound: Left ventricular ejection fraction (LVEF) ≥55%; 4) 12-leads ECG: The QT interval corrected by Fridericia method (QTcF) is less than 470 msec.
7. Voluntarily join the study and sign informed consent, with good compliance and willing to cooperate with follow-up.

Exclusion Criteria:

1. Stage IV (metastatic) breast cancer;
2. Inflammatory breast cancer;
3. There have been other malignant tumors in the past;
4. Have received anthracycline, cyclophosphamide, or anti-HER2 targeted therapy other than trastuzumab/pertuzumab;
5. Have participated in other clinical trials at the same time;
6. Have undergone major surgical procedures not related to breast cancer within 4 weeks prior to randomization or have not fully recovered from such surgical procedures;
7. Severe heart disease or discomfort, including but not limited to the following:

   History of diagnosis of heart failure or systolic dysfunction (LVEF <50%); High-risk uncontrolled arrhythmias, such as atrial tachycardia, resting heart rate> 100 bpm, significant ventricular arrhythmias (such as ventricular tachycardia) or higher-level atrioventricular block; Angina pectoris requiring antianginal medication; Clinically significant heart valve disease; ECG shows transmural myocardial infarction; Poor hypertension control (systolic blood pressure> 180 mmHg and / or diastolic blood pressure> 100 mmHg);
8. Inability to swallow, intestinal obstruction, or other factors that affect medication administration and absorption;
9. People with a known history of allergies to the drugs of this study; a history of immunodeficiency, including a positive HIV test, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
10. Pregnant and lactating female patients, female patients with fertility with baseline positive pregnancy test, or patients with fertility who are unwilling to use effective contraception during the entire trial and within 7 months after the last medication of study;
11. Suffering from a serious concomitant disease or other comorbid condition that interferes with the treatment, or any other condition that the researcher considers unsuitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
tpCR | 1 year
  the absence of invasive neoplastic cells at microscopic examination of the primary tumor and no pathological involvement of ipsilateral axillary lymph nodes at surgery

SECONDARY OUTCOMES:
Objective response rate (ORR) | 1 year
  Defined as the proportion of best overall response of either complete or partial response.
Disease free survival (DFS) | 5 years
  Defined as the time from the date of surgery to the date of recurrence/metastasis or the date of death.
3-year rate of disease-free survival | 3 years
  Defined as rate of 3-year disease-free survival
Event-free survival (EFS) | 5 years
  Defined as the time from the date of surgery to the date of recurrence/metastasis.
Number of Participants with Adverse Events | 1 year
  Defined as number of participants with adverse events related to the treatment
The quality of life | 1 year
  Using EORTC (European Organization for Research and Treatment of Cancer) QLQ-BR23 scale. The minimum and maximum values are 0 and 100, respectively. Higher scores mean better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Xu, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No